CLINICAL TRIAL: NCT00605007
Title: The Impact of Corticosteroid-induced Hyperglycemia on Clinical Outcome (Length of Stay, Disposition, APACHE Score, Need for Ventilatory Support and ICU Admission, Mortality) in Patients With COPD Exacerbation
Brief Title: Study on COPD Corticosteroid-induced Hyperglycemia on Clinical Outcome in Patients With COPD
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Principal Investigator, Emory University
Other Study IDs: IRB00001392; e1392
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2010-04

CONDITIONS: COPD
Keywords: COPD; Diabetes; Respiratory Disorders
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Diabetes Mellitus; Respiration Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Hyperglycemia is a common complication of corticosteroid (cortisone) therapy. It is estimated that more than a third of patients with chronic pulmonary disease (COPD) exacerbation (16). Despite its frequency, the impact of corticosteroid-induced diabetes on clinical outcome and mortality is not known. A computerized search of biomedical journal literature from MEDLINE, PubMed, and Ovid from 1966 to 2006 provided very little information on the prevalence and outcome of corticosteroid-induced diabetes in patients with COPD. Therefore, the present study aims to evaluate the impact of corticosteroid-induced diabetes on clinical outcome in patients with COPD exacerbation. We will perform a retrospective chart review of all patients admitted to the hospital with COPD exacerbation from 1/01/05 to 06/30/06 at Grady Memorial Hospital. Medical records of all patients with COPD exacerbation treated with corticosteroids will be analyzed. Data on demographics, laboratory values, mortality rate, rate of hypoglycemic events, length of stay, as well as disposition at discharge will be analyzed.

DETAILED DESCRIPTION:
Hypotheses:

We hypothesize that COPD patients with corticosteroid-induced hyperglycemia experience higher morbidity (infections, ventilator associated pneumonia, length of stay, acute renal failure) and mortality compared to COPD patients with normal glucose levels.

Specific Aim:

To determine the impact of corticosteroid-induced hyperglycemia on clinical outcome (length of stay, disposition, APACHE score, need for ventilatory support and ICU admission, mortality) in patients with COPD exacerbation.

ELIGIBILITY:
Inclusion Criteria: Patients admitted with COPD exacerbation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted with COPD exacerbation at Atlanta Medical Center and Grady Memorial Hospital
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2006-02; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the study is to determine the mortality rate of COPD patients with corticosteroid-induce hyperglycemia. | once all charts have been reviews

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University SOM
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States